CLINICAL TRIAL: NCT01463878
Title: Enteral Nutrition and Glycemic Variability NICU Study
Brief Title: Enteral Nutrition and Glycemic Variability Neurological Intensive Care Unit Study
Acronym: ANUS1014
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unlikely to show statistical significance and slow recruitment.
Sponsor: Eastern Virginia Medical School (Other)
Responsible Party: Principal Investigator, Paul Marik, Chief of Pulmnary and Critical Care Medicine, Eastern Virginia Medical School
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ANUS1014
Record Dates: First submitted 2011-10-24; First posted 2011-11-02 (Estimated); Results first posted 2012-09-28 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Subarachnoid Hemorrhage; Intracranial Hemorrhage; Ischemic Strokes; Subdural Hematoma
Keywords: glycemic control; glycemic variability; mean blood glucose level
MeSH Terms: conditions — Subarachnoid Hemorrhage; Intracranial Hemorrhages; Ischemic Stroke; Hematoma, Subdural

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glycerna (Experimental): Diabetic specific formula. The volume /rate of glycerna will be determined by the dietician according to standard formula.
  Interventions: Dietary Supplement: Glycerna
- Control - Jevity (Active Comparator): The control arm of the study. Patients to receive Jevity. The volume /rate of Jevity will be determined by the dietician according to standard formula.
  Interventions: Dietary Supplement: Jevity - Control Diet

INTERVENTIONS:
Dietary Supplement: Glycerna — Diabetes specific formula
  Arms: Glycerna
Dietary Supplement: Jevity - Control Diet — Control Diet
  Arms: Control - Jevity

SUMMARY:
Primary Objective:

To determine the effects of a diabetes specific enteral formula compared to a standard formula supplemented with protein (isocaloric and isonitrogenous) on the mean blood glucose and glycemic variability in a homogenous group of critically ill patients in a neurological ICU. Blood glucose will be recorded every minute using a continuous blood glucose monitor. The primary end points will be the difference between the mean blood glucose levels and the glucose variability between the control and intervention groups for the time period that the patient is in the ICU and receiving tube feeds and for up to a maximum of 14 days.

Secondary Objectives:

To determine the effects of the diabetes specific versus standard tube feeds on the change in muscle thickness and volume measured by 2-dimensional ultrasound imaging during the patients ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 89 years old
* Patients with critical illness including ischemic or hemorrhagic stroke, epidural/subdural bleeds and subarachnoid hemorrhage
* Patients who are expected to stay in the ICU for at least 5 days
* Hyperglycemia is not an inclusion criteria

Exclusion Criteria:

* Patients who have received or will be treated with systemic corticosteroids.
* Patients who will be receiving high doses of propofol (>40 cc/hr)
* Patients with type 1 Diabetes
* Patients with sepsis or acute trauma
* Patients with an expected stay in the ICU of less than 4 days
* Patients who are unable to receive enteral nutrition or who have medical conditions precluding nutrition by the enteral route including allergies to formula components
* Pregnant and lactating patients
* Patients with prior history of gastroparesis
* Patients with acute kidney failure (creatinine > 2.5mg/dl)
* Patients with acute liver failure (bilirubin > 2.0 mg/dl)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul e Marik, MD, Principal Investigator — EVMS
Locations (1):
- Sentara Norfolk General Hospital, Norfolk, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18 patients were consented and only 14 enrolled. 4 dropped out as failed to meet the inclusion criteria after consent; were bale to take food by mouth
Groups:
- Glycerna: Diabetic specific formula
- Control - Jevity: The control arm of the study. Patients to receive Jevity
Period: Overall Study
Arm/Group | Glycerna | Control - Jevity
Started | 9 | 9
Completed | 7 | 7
Not Completed | 2 | 2
Not completed — no longer met criteria for tube feed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glycerna | Control - Jevity | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 7 | 8 | 15
Age Continuous [Mean (Standard Deviation); unit: years] | 72 (12) | 74 (9) | 73 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Variability
Description: The patients blood glucose levels will be monitored with a continuous blood glucose monitor which records the calibrated blood glucose level every minute. The mean blood glucose over the patients entire ICU stay (up to 14 days) as well as the mathematical variation (fluctuation) in blood glucose levels will be calculated. The degree of glycemic variation will be assessed by a number of mathematical formula, including mean amplitude of glycemic excursions (MAGE). These parameters will be compared between the control and intervention groups.
Time Frame: Entire ICU stay. Up to 14 days in the ICU (average about 7 days)
Measure: Mean (Standard Deviation); unit: mg/dl (MAGE)
Arm/Group | Glycerna | Control - Jevity
Number analyzed (Participants) | 7 | 7
mg/dl (MAGE) | 168 (40) | 166 (41)

2. Secondary Outcome: Quadriceps Muscle Volume
Description: The quadriceps muscle volume will be estimated by 2-dimensional ultrasound imaging at enrollment and at the end of the study period (when the patient is being transferred from the ICU or no longer receiving tube feeds). The change in muscle mass during the ICU stay will be compared between the control and intervention groups.
Time Frame: First versus last measurment in ICU. Up to 14 days (average 7 days)
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Glycerna | Control - Jevity
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No